CLINICAL TRIAL: NCT05735587
Title: Dietary Intervention Targeting Inflammation, Motivation, and Engagement in Physical Activity in Sedentary, Older Adults With Depressive Symptoms
Brief Title: Blueberries, Inflammation, Motivation, and Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Courtney Millar, Assistant Scientist I, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00064749
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptoms
Keywords: Anthocyanins; Fiber; Aging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze-dried Blueberry Powder (Experimental): Randomized participants will be asked to consume 48 grams of freeze-dried blueberry powder each day for 12 weeks.
  Interventions: Other: Freeze-dried Blueberry Powder
- Placebo Powder (Placebo Comparator): Randomized participants will be asked to consume 48 grams of a nutritionally matched placebo powder devoid of fiber and anthocyanins each day for 12 weeks.
  Interventions: Other: Placebo Powder

INTERVENTIONS:
Other: Freeze-dried Blueberry Powder — Participants will be asked to consume 48 grams of freeze-dried blueberry powder (~ equivalent to 2 cups of fresh blueberries) daily for 12 weeks. Participants will be asked to save any powder packet wrappers as a means to measure compliance. They will also be instructed to avoid consumption of foods/beverages that are high in anthocyanins and/or fiber.
  Arms: Freeze-dried Blueberry Powder
Other: Placebo Powder — Participants will be asked to consume 48 grams of a nutritionally matched placebo powder (that does not contain fiber or anthocyanins) daily for 12 weeks. Participants will be asked to save any powder packet wrappers as a means to measure compliance. They will also be instructed to avoid consumption of foods/beverages that are high in anthocyanins and/or fiber.
  Arms: Placebo Powder

SUMMARY:
The purpose of this study is to determine the feasibility and preliminary efficacy of daily supplementation of freeze-dried blueberry to modulate inflammation-driven lack of motivation in 40 sedentary, older adults with depressive symptoms.

DETAILED DESCRIPTION:
The investigators will conduct a 14 week, single-site, randomized, double-blind, parallel pilot study in 40 sedentary, older adults with depressive symptoms. Participants will first enter a 2-week washout period where they will avoid consumption of foods high in fiber and anthocyanins (e.g., blueberries) and will also be wearing an activity monitor. Participants will then be randomized to consume either 48 g of freeze-dried blueberry powder (~600 mg of anthocyanins and ~8 g of fiber) or 48 g of a nutritionally matched placebo powder (devoid of anthocyanins and fiber) each day for a total of 12 weeks.

At baseline, participants will be undergo assessments for mood/well-being, relevant symptoms, motivation to engage in physical activity, and provide a blood sample for the evaluation of inflammatory biomarkers. For the entire duration of the study, participants will continue to wear the activity monitor. After 4, 6, 8 and 12 weeks of consuming the powder there will be study visits that assess mood/well-being, relevant symptoms, motivation to engage in physical activity and compliance with the intervention. Additionally, a blood sample for the evaluation of inflammatory makers will be taken after 6 and 12 weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥65 years
* Self-reporting ≥ 8 hours of sitting per/day (e.g., sedentary behavior)
* Depressive symptoms (defined as ≥4 and <16 points on the center for epidemiological studies depression-scale)

Exclusion Criteria:

* Unwilling to follow the study protocol
* A median daily step count >7,500 steps per day (as measured by the ActiGraph), or per discretion of the PI
* Cognitive impairment (defined as Montreal Cognitive Assessment, MoCA <22 points)
* Self-reporting a history of inflammatory bowel disease/syndrome, major depression, bipolar, schizophrenia, or other psychotic disorders, or per discretion of the PI
* Self-reporting type 1 or type 2 diabetes
* Allergic to intervention or control products
* Recent use (within the last 3 months) of antibiotics, or per discretion of the PI
* Recent use (within the last 3 months) of pro-biotics, or per discretion of the PI
* Current substance use disorder (Drug Abuse Screening Test, DAST-10>2 points)
* Current alcohol use disorder (Alcohol Use Disorders Identification Test - Consumption, AUDIT-C≥4 points)
* Unstable anti-depressant use (e.g., change in medication within last 3-6 months), or per discretion of the PI
* Current homicidal or suicidal ideation (assessed via the P4 Suicidality Screener)
* Current psychosis (via the Psychosis and Hallucinations Questionnaire, PHQ>12 points)
* Manic symptoms (assessed by the Mood Disorder Questionnaire, MDQ >5 points)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Millar, PhD, Principal Investigator — Hebrew SeniorLife, Marcus Institute of Aging, Harvard Medical Schools
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Millar CL, Wolfe A, Baldyga K, Dufour AB, Lipsitz LA. Berries and Steps: a protocol of a randomized, placebo-controlled pilot study testing freeze-dried blueberry powder in sedentary older adults with mild depressive symptoms. Nutr J. 2025 May 29;24(1):87. doi: 10.1186/s12937-025-01154-0. PMID 40442715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Our original goal was to recruit 40 individuals. However, recruitment was challenging and we ultimately enrolled 33 individuals. Of the 33 individuals that signed the consent form, there were 4 individuals who either did not follow the study protocol (n=2) or were lost to follow-p (n=2) before completing the baseline visit/randomization. Thus, a total of 29 individuals were enrolled and randomized.
Period: Overall Study
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Started | 15 | 14
Completed | 12 | 10
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (4) | 73 (5) | 72 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29
Height [Mean (Standard Deviation); unit: meters] | 1.6 (0.1) | 1.6 (0.1) | 1.6 (0.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 81.4 (23.0) | 80.5 (12.8) | 81.0 (18)
Median Step Count [Mean (Standard Deviation); unit: steps per day] — The median daily step count over approximately 14 days just before their baseline visit was estimated for each participant. For days that the device registered was less than 300 steps were considered missing.
  steps per day | 5916 (1257) | 6302 (1325) | 6103 (1282)
Center for Epidemiological Scale for Depression (CESD) [Mean (Standard Deviation); unit: scores on a scale] — A validated, self report questionnaire that measures of depressive symptom severity, with higher scores indicating more severe symptoms. Scores range from 0-60 points.
  scores on a scale | 8 (4) | 8 (4) | 8 (4)
Years of Education [Count of Participants; unit: Participants]
  13-15 years | 3 | 1 | 4
  16-18 years | 12 | 11 | 23
  19 or more years | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Engagement in Physical Activity
Description: Defined as change between an approximate 2-week median daily-step count prior to baseline and prior to 12 week follow-up
Time Frame: Change between baseline and 12 week follow-up
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 12 | 10
steps per day | 318 (1778) | 346 (624)

2. Secondary Outcome: Study Recruitment Feasibility
Description: Participant retention (e.g., the number of participants that complete the intervention out of all participants randomized to an intervention arm)
Time Frame: Through study completion, approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 15 | 14
Participants | 12 | 10

3. Secondary Outcome: Change in Motivation
Description: Motivation to engage in physical activity will be assessed via self-report questionnaire, Motives for Physical Activities Measure-Revised (range 0-30 points, with higher scores indicating higher levels of motivation).
Time Frame: Change between baseline and 12 week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 12 | 10
score on a scale | 4 (18) | 0 (12)

4. Secondary Outcome: Change in Inflammatory Marker - C-Reactive Protein
Description: C-reactive protein (mg/L) will be measured in blood collected from participants.
Time Frame: Change between Baseline and 12 week follow-up.
Measure: Mean (Standard Deviation); unit: miligrams/liter
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 12 | 10
miligrams/liter | 0.6 (2.6) | -1.6 (4.9)

5. Secondary Outcome: Change in Inflammatory Marker - Interleukin-6
Description: Interleukin-6 (pg/mL) will be measured in blood collected from participants. If values were above the standard curve in the ELISA kit (n= 2 samples), then the highest standard concentration was used as the value.
Time Frame: Change between Baseline and 12 week follow-up
Measure: Mean (Standard Deviation); unit: picograms/mililiter
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 12 | 10
picograms/mililiter | -0.5 (1.2) | -0.7 (2.6)

6. Secondary Outcome: Change in Inflammatory Marker - Brain Derived Neurotrophic Factor
Description: Brain derived neurotrophic (ng/mL) factor will be measured in blood collected from participants.
Time Frame: Change between Baseline and 12 week follow-up
Measure: Mean (Standard Deviation); unit: nanograms/mL
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 12 | 10
nanograms/mL | 1.258 (10.038) | -1.226 (12.116)

ADVERSE EVENTS:
Time Frame: Adverse events were captured throughout the study duration of each participant, which was approximately 14 weeks.
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 4/15 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Freeze-dried Blueberry Powder (N=15) | Placebo Powder (N=14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased frequency of bowel movements (Gastrointestinal disorders) | 1 (1) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Unpleasant taste and/or experience while taking study powder (Product Issues) | 0 (0) | 2 (2) — Described as "a lingering blueberry taste" or as an "irritated esophagus"
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
High Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1) — This occurred at baseline. Participant was aware this issue was present prior to our study and had been trying to get an appointment with their doctor. Study staff contacted their doctor and the participant was received treatment.
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05735587/Prot_SAP_001.pdf